CLINICAL TRIAL: NCT05263453
Title: A Single-arm, Multi-center Phase II Trial to Evaluate the Efficacy and Safety of the Combination of HL-085 and Vemurafenib in Advanced Melanoma Patients With BRAF V600E/K Mutation
Brief Title: HL-085+Vemurafenib to Treat Advanced Melanoma Patients With BRAF V600E/K Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-102-II-01
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HL-085+Vemurafenib (Experimental): HL-085 12mg BID+Vemurafenib 720mg BID combination therapy
  Interventions: Drug: HL-085; Drug: Vemurafenib

INTERVENTIONS:
Drug: HL-085 — HL-085 capsule 12mg administered orally twice daily in a 21-day treatment cycle
Drug: Vemurafenib — Vemurafenib tablet 720mg administered orally twice daily in a 21-day treatment cycle

SUMMARY:
The main purpose of this study is to Evaluate the Efficacy and Safety of the combination of HL-085 and Vemurafenib in Advanced Melanoma Patients with BRAF V600E/K Mutation. This study includes IIa and IIb phase. Phase IIa will determine the dose regiment for Phase IIb. Phase IIb part will evaluate the efficacy and safety with this combination regiment.

DETAILED DESCRIPTION:
This is a single-arm, multi-center Phase II trial to evaluate the efficacy and safety of the combination of HL-085 and Vemurafenib in advanced melanoma patients with BRAF V600E/K mutation. There are two phase of this study ( IIa and IIb). Phase IIa will be evaluating the safety and efficacy of the combination regiment (HL-08512mg +Vemurafenib 720mg, and/or some lower dose regiment, such as 9mg+720mg) in 20-30 patients, and final determine the recommended dose regiment for Phase IIb. In Phase IIb will enrolled 74 patients , the primary endpoint is ORR, and the secondary endpoint are PFS. The safety profile of this combined HL-085/Vemurafenib regimen will be monitored during both phases. The treatment period consists of 21-day cycles until progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age;
* Patients with histological confirmed advanced melanoma;
* BRAF V600E/ V600K mutation positive；
* At least 1 site of radiographically measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status(PS) of 0 to 1;
* Life expectancy ≥ 3 months;
* Can swallow the medicine,
* UCG documenting LVEF ≥50% within seven days prior to initiation of dosing;
* Adequate hematologic, renal, and liver function as defined by laboratory values performed within 42 days prior to initiation of dosing: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelet count ≥ 1.0 x lower limit of normal (LLN); Hemoglobin ≥ 90 g/L; Serum creatinine ≤ 1.5 x upper limit of normal (ULN); Serum aspartate transaminase (AST) or serum alanine transaminase (ALT)≤ 2.5x ULN, and ≤ 5.0 x ULN if liver metastases are present. Serum alkaline phosphatase （ALP）≤ 2.5x ULN and ≥ 2.5 x ULN if bone metastases are present; Total serum bilirubin ≤ 1.5 x ULN; Serum albumin ≥ 30 g/L; Coagulation function：INR ≤1.5×ULN；Activated partial thrombin time (APTT) ≤1.5×ULN; Creatine kinase (CK) ≤1× ULN
* 10. Before study entry, written informed consent must be obtained from the patient prior to performing any study-related procedures.
* 11. Be willing and able to complete all the study procedures and follow-up examinations.

Exclusion Criteria:

* Patients who have been previously treated with a BRAF and/or MEK inhibitors.
* Patients with active CNS lesions are excluded (i.e. those with radiographically unstable, symptomatic lesions). However, patients treated with stereotactic therapy or surgeries are eligible if patient remains without evidence of disease progression in brain ≥ 3 months.
* Patients accepted other administration of anti-cancer study therapies within 4 weeks prior to initiation of dosing;
* Dysphagia，refractory nausea, vomiting, small bowel resection or any other gastrointestinal ailment that would preclude study drug absorption.
* Major surgery or traumatic injury (exclude baseline biopsy ) within 14 days prior to first dose of study treatment
* Patients have mean QTcB interval ≥ 480 msec, or any history of congenital long QT syndrome or with ongoing concomitant treatment with medications that prolong the QT interval at screening;
* Serious illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, uncontrolled hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, symptomatic autoimmune diseases, severe obstructive or restrictive pulmonary diseases, uncontrolled endocrine disorders (hypothyroidism, hyperthyroidism and diabetes mellitus), retinopathy, active systemic infections, and inflammatory bowel disorders. This includes known HIV or AIDS-related illness, or active HBV and HCV.
* Active infection or antibiotics within one-week prior to study, including unexplained fever
* Lactating females or pregnant females.
* Systemic steroid or other immunosuppressive therapy within 4 weeks of starting the study.
* Any significant psychiatric disease, medical intervention, or other condition, which in the opinion of the principal investigator, could prevent adequate informed consent or compromise participation in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
  Objective response rate (ORR)as measure of efficacy by RECIST 1.1

SECONDARY OUTCOMES:
Progression Free survival （PFS） | up to 24 months
  Defined as the time from first dosing (C1D1) to date of first observed progression or death from any cause (whichever comes first)
Disease control rate（DCR） | up to 24 months
  Defined as the percentage of patients who have achieved a confirmed response of at least CR or PR or a response of SD

OTHER OUTCOMES:
Grade 3, 4, 5 toxicities | up to 24 months
  Reporting of all grade 3, 4, 5 toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, Ph.D, Study Chair — Shanghai Kechow Pharma, Inc.
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided